CLINICAL TRIAL: NCT07082842
Title: A Multicenter, Parallel, Randomized, Placebo (Double-blind) and Pirfenidone (Open-label) Controlled Phase III Clinical Trial Evaluating the Efficacy and Safety of HEC585 Tablets in Patients With Idiopathic Pulmonary Fibrosis (IPF)
Brief Title: Confirmatory Clinical Study of HEC585 Tablets in Patients With IPF
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sunshine Lake Pharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HEC585-IPF-301
Record Dates: First submitted 2025-07-02; First posted 2025-07-24 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Idiopathic Pulmonary Fibrosis (IPF)
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis | interventions — pirfenidone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- HEC585 (Experimental)
  Interventions: Drug: HEC585
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- pirfenidone (Active Comparator)
  Interventions: Drug: Pirfenidone

INTERVENTIONS:
Drug: HEC585 — HEC585 tablet, taken once daily
  Arms: HEC585
Drug: Placebo — HEC585 Simulation Board, taken once daily
  Arms: Placebo
Drug: Pirfenidone — Pirfenidone, taken three times a day
  Arms: pirfenidone

SUMMARY:
A multicenter, parallel, randomized, placebo (double-blind) and pirfenidone (open-label) controlled Phase III clinical trial to evaluate the efficacy and safety of HEC585 in patients with idiopathic pulmonary fibrosis (IPF)

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily participate in this clinical study and sign the informed consent form before the study begins;
2. When signing the informed consent form, the age should be between 40 and 80 years old (inclusive of 40 and 80), and gender is not restricted;
3. Be diagnosed with IPF according to the diagnostic criteria of the IPF clinical practice guidelines jointly released by the American Thoracic Society, the European Respiratory Society, the Japanese Respiratory Society and the Latin American Thoracic Society in 2022 ; Chest high-resolution computed tomography (HRCT) examination (HRCT examination within 3 months before screening) or lung biopsy (if any) should be confirmed by central reading;
4. The ratio of forced expiratory volume in one second (FEV1) to forced vital capacity (FVC) at the screening period is ≥ 0.7;
5. The percentage of FVC as a percentage of the normal predicted value at the screening period is ≥ 45%;
6. The percentage of DLco (hemoglobin [Hb] corrected) as a percentage of the normal predicted value at the screening period is ≥ 30%;
7. Female or male subjects with potential fertility agree and commit to taking effective contraceptive measures from the time of signing the informed consent form until 30 days after the last administration of the investigational drug; at the same time, avoid sperm/egg collection, sperm/egg donation;
8. According to the assessment by the investigator, the subjects are willing and able to comply with the requirements of the protocol and attend the visits.

Exclusion Criteria:

1. The researchers believe that the subjects experienced significant deterioration of IPF within the first three months of the randomization period.
2. Other known causes of interstitial lung disease, such as exposure to the home or occupational environment, connective tissue diseases, drug toxicity, etc.
3. Abnormalities in the lungs or chest that are clinically significant and judged by the researchers to potentially affect the trial results.
4. Within one month before randomization, any active infection requiring systemic treatment (such as oral or intravenous administration) in the form of activity (including bacterial, viral, parasitic or fungal infections).
5. Expected to undergo lung transplantation during the course of the study.
6. Expected survival period less than 6 months.
7. History of malignant tumors within the previous 5 years (excluding localized cancers such as basal cell carcinoma).
8. Moderate to severe liver dysfunction (Child-Pugh classification of grade B or C).
9. Within six months before screening, history of unstable or deteriorating heart disease, including but not limited to the following conditions:

   1. Unstable angina pectoris;
   2. Myocardial infarction;
   3. Congestive heart failure requiring hospitalization or NYHA III/IV grade;
   4. Uncontrolled severe arrhythmia.
10. Unable to perform the 6MWT or pulmonary function test, such as if the patient is mentally unstable and unable to cooperate, etc.;
11. Allergic to any component of Ifinonate Hydrochloride Tablets (except the active ingredient, the excipients include microcrystalline cellulose, pre-gelatinized starch, cross-linked povidone, povidone, dibutyl hydroxytoluene, colloidal silicon dioxide, magnesium stearate, polyvinyl alcohol, polyethylene glycol, talc and titanium dioxide) or pirfenidone tablets;
12. The last administration of the study drug for other clinical trials occurred within 4 weeks before randomization or 5 half-lives (whichever is longer);
13. Pregnant or breastfeeding;
14. Within 3 months before screening, had a smoking history or was unwilling to maintain a smoking-free status during the study;
15. Within 6 months before screening, frequently drank alcohol [average weekly alcohol consumption exceeding 21 units (1 unit = 360 mL of beer, or 150 mL of wine, or 45 mL of 40% alcohol spirits)];
16. Had a history of drug abuse within 6 months before screening;
17. Has a family or personal history of long QT interval syndrome;
18. The investigator believes that the subject has conditions that may compromise their safety or compliance, significantly affect the pharmacokinetics of the drug, or prevent them from completing the study.
19. During the screening period, liver function test values exceeded any of the following standards: total bilirubin > 1.5 times the upper limit of normal (ULN); aspartate aminotransferase or alanine aminotransferase > 2 times ULN;
20. During the screening period, glomerular filtration rate < 45 mL/min/1.73 m2, calculated using the CKD-EPI (based on serum creatinine) formula ;
21. At the time of screening, human immunodeficiency virus antibody or syphilis spirochete antibody test results were positive;
22. At the time of screening, there was an uncontrolled hepatitis B virus infection (positive hepatitis B surface antigen, and hepatitis B DNA ≥ 2x102 IU/mL) or hepatitis C virus infection (positive anti-hepatitis C antibody and hepatitis C RNA);
23. During the screening period, QTcF > 480 ms (using the Fridericia formula, QTcF = QT/RR^0.33).
24. Those who have previously taken isoniazidine hydrochloride;
25. Within the first 4 weeks before randomization, used any of the following treatments:

    1. Any cytotoxic drugs or immunosuppressants, including but not limited to azathioprine, cyclophosphamide, methotrexate, cyclosporine, etc.;
    2. Pirfenidone or nintedanib;
    3. > 15 mg/d prednisone or equivalent dose of other glucocorticoids;
    4. Strong inducers or inhibitors of CYP3A4, CYP2C8 or CYP2C19 (including but not limited to ritonavir, clarithromycin, aletris, carbamazepine, gemfibrozil, fluoxetine, fluvoxamine, etc.);
    5. Moderate, strong inhibitors or inducers of CYP1A2 (including but not limited to fluvoxamine, ciprofloxacin, enoxacin, etc.).

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 472 (Estimated)
Dates: Start 2025-10-09 (Estimated); Primary Completion 2031-01-15 (Estimated); Study Completion 2032-02-15 (Estimated)

PRIMARY OUTCOMES:
Change in FVC from baseline at 52 weeks (mL) | 52week

SECONDARY OUTCOMES:
The interval (in days) from the start of the study until the first occurrence of any of the following clinical events (whichever occurs first) within 52 weeks | 52week
The percentage of FVC relative to the predicted value (%FVC) compared to the baseline value changes | 52week
The percentage of DLco(Hb-correction) relative to the expected value [%DLco(Hb-correction)] and the change from the baseline value | 52week
The total walking distance of 6MWT（six minutes walk ）test compared to the baseline value | 52week
  The longer the 6MWT distance is, the better the patient's disease condition is.
The change in SGRQ（St George's Respiratory Questionnaire） score compared to the baseline | 52week
  A lower SGRQ score indicates a better disease condition for the subject.

IPD SHARING:
Plan to Share IPD: No